CLINICAL TRIAL: NCT01670578
Title: Platelet-rich Plasma (PRP) vs Viscosupplementation in the Treatment of Knee Articular Degenerative Pathology: a Randomized Double-blind Controlled Trial
Brief Title: Platelet-rich Plasma vs Viscosupplementation in the Treatment of Knee Articular Degenerative Pathology
Acronym: PRP2009
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KNEEJECT
Record Dates: First submitted 2012-08-13; First posted 2012-08-22 (Estimated); Last update posted 2017-10-30 (Actual); Status verified 2017-10

CONDITIONS: Knee Chondropathy; Osteoarthritis, Knee
Keywords: P.R.P.; viscosupplementation; double-blind randomized; intra-articular injections; knee degenerative pathology; early osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PRP Group (Experimental): Patients (n=96) randomized to this group of treatment will receive 3 blinded knee intra-articular injections of autologous Platelet-Rich Plasma one week apart each other.
  Interventions: Biological: PRP
- Hyaluronan Group (Active Comparator): Patients (n=96) randomized to this group of treatment will receive 3 blinded knee intra-articular injections of hyaluronic acid ( Hyalubrix 30 mg/2ml, Fidia Farmaceutici Spa, Italy) one week apart each other.
  Interventions: Device: Hyaluronic acid

INTERVENTIONS:
Biological: PRP
  Arms: PRP Group
Device: Hyaluronic acid
  Other Names: Hyalubrix fl. 30 mg/2ml, Fidia farmaceutici Spa, Italy
  Arms: Hyaluronan Group

SUMMARY:
The investigators hypothesized that intra-articular injections of Platelet-rich Plasma (PRP) to treat knee degenerative articular cartilage pathology could determine pain relief and recovery of knee function with overall clinical outcome comparable or even better than viscosupplementation, which is a common injective approach applied in this kind of pathology. To this purpose the investigators designed a double blind randomized controlled trial comparing PRP vs viscosupplementation.

A power analysis has been performed for the primary endpoint of IKDC (International Knee Documentation Committee) subjective score improvement at the 12-month follow-up for PRP. From a pilot study, a standard deviation of 15.2 points was found. With an alpha error of 0.05, a beta error of 0.2 and a minimal clinically significant difference of 6.7 points corresponding at 1/3 of the documented mean improvement, the minimum sample size was 83 for each group. Considering a possible drop out of 15%, 96 patients per group are required for total 192 patients, selected according to well-defined inclusion criteria (see 'Eligibility criteria' section). Patients are then assigned to two different treatment groups, according to a randomization list. The first group of treatment consists of three weekly intra-articular injections of autologous PRP obtained with the following procedure: a 150-ml autologous venous blood sample undergoes 2 centrifugations (the first at 1480 rpm for 6 minutes to separate erythrocytes, and a second at 3400 rpm for 15 minutes to concentrate platelets) to produced 20 ml of PRP. This unit of PRP is then divided into 4 small units of 5 ml each. One unit is sent to the laboratory for analysis of platelet concentration and for a quality test, 3 units are stored at -30° C.

The second treatment group consists of patients receiving three weekly injections of hyaluronic acid (Hyalubrix 30 mg/2ml, Fidia Farmaceutici Spa, Italy;Molecular Weight: 1500 kDa).

To guarantee the blinding of the patients, all of them undergo blood harvesting to obtain autologous PRP which will be used only in half of them, according to the aforementioned randomization list. One week after the PRP production, the injective treatment starts, with 3 weekly injections of PRP or HA. At the moment of the injection the syringe is properly covered to prevent the patient from discovering the substance he was receiving. After the injection, patients are sent home with instructions to limit the use of the leg for at least 24 h and to use cold therapy/ice on the affected area to relieve pain. During this period, the use of non-steroidal medication is forbidden.

Patients are prospectively evaluated basally and at 2, 6, and 12 months of follow-up using clinical subjective scores and objective parameters to determine clinical outcome (see 'Outcome measure' section). Patient satisfaction and adverse events will be also reported. All the clinical evaluations are performed by a medical staff not involved in the injective procedure, in order to keep the study double blinded. At the end of the study, the nature of the injected substance is revealed to the patients.

DETAILED DESCRIPTION:
Current research is investigating new methods for stimulating repair or replacing damaged cartilage. In particular, the most recent knowledge regarding tissue biology highlights a complex regulation of growth factors (GFs) for the normal tissue structure and the reaction to tissue damage. The influence of GFs on cartilage repair is now widely investigated in vitro and in vivo. Platelet Rich Plasma (PRP) is a simple, low- cost and minimally- invasive method that allows one to obtain a natural concentrate of autologous GFs from the blood, and it is increasingly applied in the clinical practice to treat knee degenerative pathology, such as chondropathy and early osteoarthritis (OA). The biological rational of PRP is that platelets contain storage pools of GFs, cytokines, chemokines and many other mediators.Although its widespread application, there are no high level studies in the literature to demonstrate the real efficacy of PRP. In fact, at the present moment, to our knowledge there is no published randomized controlled trial comparing PRP with other conservative treatments commonly used for knee OA.

The investigators hypothesized that intra-articular injections of PRP to treat knee degenerative articular cartilage pathology could determine pain relief and recovery of knee function with overall clinical outcome comparable or even better than viscosupplementation, which is a common injective approach applied in this kind of pathology. To this purpose the investigators designed a double blind randomized controlled trial comparing PRP vs viscosupplementation.

A power analysis has been performed for the primary endpoint of IKDC subjective score improvement at the 12-month follow-up for PRP. From a pilot study, a standard deviation of 15.2 points was found. With an alpha error of 0.05, a beta error of 0.2 and a minimal clinically significant difference of 6.7 points corresponding at 1/3 of the documented mean improvement, the minimum sample size was 83 for each group. Considering a possible drop out of 15%, 96 patients per group are required for total 192 patients. Patients are then assigned to two different treatment groups, according to a randomization list. The first group of treatment consists of three weekly intra-articular injections of autologous PRP obtained with the following procedure: a 150-ml autologous venous blood sample undergoes 2 centrifugations (the first at 1480 rpm for 6 minutes to separate erythrocytes, and a second at 3400 rpm for 15 minutes to concentrate platelets) to produced 20 ml of PRP. This unit of PRP is then divided into 4 small units of 5 ml each. One unit is sent to the laboratory for analysis of platelet concentration and for a quality test, 3 units are stored at -30° C.

The second treatment group consists of patients receiving three weekly injections of hyaluronic acid (Hyalubrix 30 mg/2ml, Fidia Farmaceutici Spa, Italy;Molecular Weight: 1500 kDa).

To guarantee the blinding of the patients, all of them undergo blood harvesting to obtain autologous PRP which will be used only in half of them, according to the aforementioned randomization list. One week after the PRP production, the injective treatment starts, with 3 weekly injections of PRP or HA. At the moment of the injection the syringe is properly covered to prevent the patient from discovering the substance he was receiving. After the injection, patients are sent home with instructions to limit the use of the leg for at least 24 h and to use cold therapy/ice on the affected area to relieve pain. During this period, the use of non-steroidal medication is forbidden.

Furthermore, at the moment of each weekly injection, before injecting the substance, an attempt of harvesting synovial fluid is performed. During the same visit, also a peripheral blood sample (3 ml) is taken. These samples are then sent to a dedicated Laboratory in order to test the concentration of some GFs, pro and anti-inflammatory cytokines, both at local (synovial fluid) and systemic level (peripheral blood). The aim is to evaluate the trend in the concentration rate of these molecules over the period of the injective treatment.

Patients are prospectively evaluated basally and at 2, 6, and 12 months of follow-up using IKDC, KOOS (Knee Injury and Osteoarthritis Outcome Score), EQ-VAS (Visual Analogue Scale) for general health status, and Tegner scores. Furthermore at basal evaluation and at every follow-up the ROM (Range of Motion) and the transpatellar circumference of both the index knee and the contralateral one are measured to check if any changes occurred over time. Patient satisfaction and adverse events will be also reported.

During follow-up evaluations, also a peripheral blood sample is harvested (as described before) in order to assess any eventual variation in the concentration of same GFs, pro and anti-inflammatory cytokines previously evaluated. All the clinical evaluations are performed by a medical staff not involved in the injective procedure, in order to keep the study double blinded. At the end of the study, the nature of the injected substance is revealed to the patients.

ELIGIBILITY:
Inclusion Criteria:

* patients affected by knee articular degenerative pathology with history of chronic (for at least 4 months) pain or swelling;
* imaging findings of degenerative changes of the joint (Kellgren Lawrence 0 to III at X-ray evaluation).

Exclusion Criteria:

* age > 80 years;
* Kellgren-Lawrence score at X-ray evaluation > 3;
* major axial deviation (varus >5° , valgus > 5°),
* systemic disorders such as diabetes, rheumatoid arthritis, haematological diseases (coagulopathy), severe cardiovascular diseases, infections, immunodepression;
* patients in therapy with anticoagulants or antiaggregants;
* use of NSAIDs in the 5 days before blood donation;
* patients with Hb values < 11 g/dl and platelet values < 150,000/mmc.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2009-02; Primary Completion 2013-08 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
IKDC (International Knee Documentation Committee) subjective score variation for both groups of treatment at 12 months of follow-up (f-up) | baseline and 12 months of follow-up

SECONDARY OUTCOMES:
IKDC (International Knee Documentation Committee) subjective score variation for both groups of treatment at 6 months of follow-up (f-up) | baseline and 6 months of follow-up
IKDC (International Knee Documentation Committee) subjective score variation for both groups of treatment at 2 months of follow-up (f-up) | baseline and 2 months of follow-up
IKDC (International Knee Documentation Committee) objective score variation for both groups of treatment at 12 months of follow-up (f-up) | baseline and 12 months of follow-up
IKDC (International Knee Documentation Committee) objective score variation for both groups of treatment at 6 months of follow-up (f-up) | baseline and 6 months of follow-up
IKDC (International Knee Documentation Committee) objective score variation for both groups of treatment at 2 months of follow-up (f-up) | baseline and 2 months of follow-up
VAS (Visual Analogue scale) for General Health Status variation for both groups of treatment at 12 months of follow-up (f-up) | baseline and 12 months of follow-up
VAS (Visual Analogue scale) for General Health Status variation for both groups of treatment at 6 months of follow-up (f-up) | baseline and 6 months of follow-up
VAS (Visual Analogue scale) for General Health Status variation for both groups of treatment at 2 months of follow-up (f-up) | baseline and 2 months of follow-up
Tegner score variation for both groups of treatment at 12 months of follow-up (f-up) | baseline and 12 months of follow-up
Tegner score variation for both groups of treatment at 6 months of follow-up (f-up) | baseline and 6 months of follow-up
Tegner score variation for both groups of treatment at 2 months of follow-up (f-up) | baseline and 2 months of follow-up
KOOS (Knee injury and Osteoarthritis Outcome Score) variation for both groups of treatment at 12 months of follow-up (f-up) | baseline and 12 months of follow-up
KOOS (Knee injury and Osteoarthritis Outcome Score) variation for both groups of treatment at 6 months of follow-up (f-up) | baseline and 6 months of follow-up
KOOS (Knee injury and Osteoarthritis Outcome Score) variation for both groups of treatment at 2 months of follow-up (f-up) | baseline and 2 months of follow-up
Knee Range of Motion (ROM) variation for both groups of treatment at 12 months of follow-up (f-up) | baseline and 12 months of follow-up
  Every patient had both knees' ROM measured to eventually assess any variation between the treated and un-treated knee during the follow-up evaluation
Knee Range of Motion variation for both groups of treatment at 6 months of follow-up (f-up) | baseline and 6 months of follow-up
Knee Range of Motion variation for both groups of treatment at 2 months of follow-up (f-up) | baseline and 2 months of follow-up
Knee Trans patellar and distal quadriceps circumference variation for both groups of treatment at 12 months of follow-up (f-up) | baseline and 12 months of follow-up
Knee Trans patellar and distal quadriceps circumference variation for both groups of treatment at 6 months of follow-up (f-up) | baseline and 6 months of follow-up
Knee Trans patellar and distal quadriceps circumference variation for both groups of treatment at 2 months of follow-up (f-up) | baseline and 2 months of follow-up
Patient global satisfaction for the treatment | 12 months
Pain Level on a Visual Analogue Score after each intra-articular injection | 7 days after each injection
Swelling Level on a Visual Analogue Score after each injection | 7 days after each injection
Number of Participants with Adverse Events | 2, 6, 12 months of follow up
  Type, duration and trend of every adverse event for each patient will be reported
Pain Duration after each intra-articular injection | 7 days after each injection
Swelling Duration after each injection | 7 days after each injection
Trend in the concentration of GFs and cytokines in synovial fluid | Baseline, day 7 (second injection), day 14 (third injection)
Trend in the concentration of GFs and cytokines in peripheral blood | Baseline, day 7 (second injection), day 14 (third injection), 2 months, 6 months, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Elizaveta Kon, MD, Principal Investigator — III Orthopaedic Clinic and Nano-biotechnology Lab, Rizzoli Orthopaedic Institute, Bologna, Italy
Locations (1):
- III Orthopaedic Clinic and Nano-biotechnology Lab, Rizzoli Orthopaedic Institute, Bologna, Emilia-Romagna, Italy

REFERENCES:
- [Background] Sanchez M, Azofra J, Anitua E, Andia I, Padilla S, Santisteban J, Mujika I. Plasma rich in growth factors to treat an articular cartilage avulsion: a case report. Med Sci Sports Exerc. 2003 Oct;35(10):1648-52. doi: 10.1249/01.MSS.0000089344.44434.50. PMID 14523300
- [Background] Everts PA, Knape JT, Weibrich G, Schonberger JP, Hoffmann J, Overdevest EP, Box HA, van Zundert A. Platelet-rich plasma and platelet gel: a review. J Extra Corpor Technol. 2006 Jun;38(2):174-87. PMID 16921694
- [Background] Tschon M, Fini M, Giardino R, Filardo G, Dallari D, Torricelli P, Martini L, Giavaresi G, Kon E, Maltarello MC, Nicolini A, Carpi A. Lights and shadows concerning platelet products for musculoskeletal regeneration. Front Biosci (Elite Ed). 2011 Jan 1;3(1):96-107. doi: 10.2741/e224. PMID 21196289
- [Background] Grimaud E, Heymann D, Redini F. Recent advances in TGF-beta effects on chondrocyte metabolism. Potential therapeutic roles of TGF-beta in cartilage disorders. Cytokine Growth Factor Rev. 2002 Jun;13(3):241-57. doi: 10.1016/s1359-6101(02)00004-7. PMID 12486877
- [Background] Sanchez AR, Sheridan PJ, Kupp LI. Is platelet-rich plasma the perfect enhancement factor? A current review. Int J Oral Maxillofac Implants. 2003 Jan-Feb;18(1):93-103. PMID 12608674
- [Background] Hickey DG, Frenkel SR, Di Cesare PE. Clinical applications of growth factors for articular cartilage repair. Am J Orthop (Belle Mead NJ). 2003 Feb;32(2):70-6. PMID 12602635
- [Background] Sampson S, Reed M, Silvers H, Meng M, Mandelbaum B. Injection of platelet-rich plasma in patients with primary and secondary knee osteoarthritis: a pilot study. Am J Phys Med Rehabil. 2010 Dec;89(12):961-9. doi: 10.1097/PHM.0b013e3181fc7edf. PMID 21403592
- [Background] Wang-Saegusa A, Cugat R, Ares O, Seijas R, Cusco X, Garcia-Balletbo M. Infiltration of plasma rich in growth factors for osteoarthritis of the knee short-term effects on function and quality of life. Arch Orthop Trauma Surg. 2011 Mar;131(3):311-7. doi: 10.1007/s00402-010-1167-3. Epub 2010 Aug 17. PMID 20714903
- [Background] Kon E, Filardo G, Di Martino A, Marcacci M. Platelet-rich plasma (PRP) to treat sports injuries: evidence to support its use. Knee Surg Sports Traumatol Arthrosc. 2011 Apr;19(4):516-27. doi: 10.1007/s00167-010-1306-y. Epub 2010 Nov 17. PMID 21082164
- [Background] Kon E, Buda R, Filardo G, Di Martino A, Timoncini A, Cenacchi A, Fornasari PM, Giannini S, Marcacci M. Platelet-rich plasma: intra-articular knee injections produced favorable results on degenerative cartilage lesions. Knee Surg Sports Traumatol Arthrosc. 2010 Apr;18(4):472-9. doi: 10.1007/s00167-009-0940-8. Epub 2009 Oct 17. PMID 19838676
- [Background] Filardo G, Kon E, Buda R, Timoncini A, Di Martino A, Cenacchi A, Fornasari PM, Giannini S, Marcacci M. Platelet-rich plasma intra-articular knee injections for the treatment of degenerative cartilage lesions and osteoarthritis. Knee Surg Sports Traumatol Arthrosc. 2011 Apr;19(4):528-35. doi: 10.1007/s00167-010-1238-6. Epub 2010 Aug 26. PMID 20740273
- [Derived] Di Martino A, Di Matteo B, Papio T, Tentoni F, Selleri F, Cenacchi A, Kon E, Filardo G. Platelet-Rich Plasma Versus Hyaluronic Acid Injections for the Treatment of Knee Osteoarthritis: Results at 5 Years of a Double-Blind, Randomized Controlled Trial. Am J Sports Med. 2019 Feb;47(2):347-354. doi: 10.1177/0363546518814532. Epub 2018 Dec 13. PMID 30545242